CLINICAL TRIAL: NCT05550480
Title: Effect of Continuous Glucose Monitoring on Hypoglycemia in Adults With Pancreatogenic Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Soren Schou Olesen, Professor, Chief Physician, MD, PhD, Aalborg University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: N-20210064; N-20210064 (Other: North Denmark Region Committee in Health Research Ethics)
Record Dates: First submitted 2022-09-15; First posted 2022-09-22 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Pancreatogenic Type 3C Diabetes Mellitus
Keywords: Chronic pancreatitis; Pancreatic Diseases; Digestive System Diseases; Diabetes; Continuous Glucose Monitoring
MeSH Terms: conditions — Pancreatitis, Chronic; Pancreatic Diseases; Digestive System Diseases; Diabetes Mellitus | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continuous glucose monitoring (Experimental): Participants will monitor their glucose levels using CGM with access to interstitial glucose levels continuously throughout the day.
  Each study period is preceded by 20 days of masked CGM assessment.
  Interventions: Device: Continuous glucose monitoring
- Self-monitoring of blood glucose (No Intervention): Participants will monitor their blood glucose levels using a glucometer and a capillary blood sample from finger-pricking. Participants will in addition use masked CGM for the last 20 days of the study period to monitor glucose levels for comparison.
  Each study period is preceded by 20 days of masked CGM assessment.

INTERVENTIONS:
Device: Continuous glucose monitoring — Continuous glucose monitoring for 50 days
  Other Names: CGM
  Arms: Continuous glucose monitoring

SUMMARY:
This study will investigate the effect of continuous glucose monitoring (CGM) (compared to self-monitoring) on hypoglycemia and glycemic control in patients with insulin-treated pancreatogenic diabetes.

DETAILED DESCRIPTION:
The use of CGM in people with type 1 or type 2 diabetes receiving multiple daily insulin injections improves glycemic control and reduces time spent in hypoglycemia compared to self-monitoring. These beneficial effects of CGM are likely also present in people with pancreatogenic diabetes but have only been sparsely investigated.

In this study, the investigators, therefore, aim to investigate the effects of CGM (compared to self-monitoring) on hypoglycemia and glycemic control in patients with pancreatogenic diabetes. Patients with chronic pancreatitis and insulin-treated diabetes will be randomized 1:1 to receive 50 days of CGM followed by 50 days of self-monitoring or vice versa. Each study period is preceded by 20 days of masked CGM assessment, which also serves as the washout period between the two study periods. Furthermore, the self-monitoring group will use masked CGM for the last 20 days of the study period to monitor glucose levels for comparison with the unmasked CGM period. Thus, each study period lasts a total of 70 days.

The investigators hypothesize that the use of CGM vs self-monitoring of blood glucose in patients with pancreatogenic diabetes will lead to decreased time spent with a glucose value <3.0 mmol/l and increased time in glycemic range.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent before any study specific procedures
* Able to read and understand Danish
* Male or female age ≥ 18 ≤ 85 years
* A definitive diagnosis of chronic pancreatitis based on the M-ANNHEIM criteria
* A diagnosis of insulin treated pancreatogenic diabetes based on the World Health Organization criteria for diabetes (HbA1c ≥6.5 % (48 mmol/mol) and/or fasting plasma glucose ≥126 mg/dl (7.0 mmol/l)) >3 months after diagnosis of pancreatitis

Exclusion Criteria:

* Known or suspected abdominal cancer (incl. intestine, pancreas, and the hepato-biliary system)
* Severe pre-existing comorbidities (assessed by investigator upon inclusion)
* Attack of acute on chronic pancreatitis requiring admission within four weeks prior to inclusion
* Use of glucocorticoid medications within four weeks prior to inclusion, with the exception of inhaled glucocorticoids in the treatment of chronic pulmonary diseases.
* Presence of autoimmune antibodies suggestive of type 1 diabetes
* Prior pancreatic surgery (including total pancreatectomy, pancreaticoduodenectomy, distal pancreatectomy, pancreaticojejunostomy, enucleation, or Frey procedure)
* Prior gastric surgery or vagotomy
* Autoimmune pancreatitis

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-09-08 (Actual); Primary Completion 2024-06-05 (Actual); Study Completion 2024-06-05 (Actual)

PRIMARY OUTCOMES:
Time spent with glucose value <3.0 mmol/l (level 2 hypoglycemia) | In period 1, the observation period begins on day 50 ±2 days of the study and ends on day 70 ±2 days. In period 2, the observation period starts on day 120 ±2 days and ends on day 140 ±2 days.
  The difference between CGM and self-monitoring of blood glucose in time spent with glucose value <3.0 mmol/l (level 2 hypoglycemia) measured by CGM.

SECONDARY OUTCOMES:
Time in range (glucose value 3.9 - 10.0 mmol/l) | In period 1, the observation period begins on day 50 ±2 days of the study and ends on day 70 ±2 days. In period 2, the observation period starts on day 120 ±2 days and ends on day 140 ±2 days.
  The difference between CGM and self-monitoring of blood glucose in time in range (glucose value 3.9 - 10.0 mmol/L) measured by CGM.
Time below range (glucose <3.9 mmol/L) | In period 1, the observation period begins on day 50 ±2 days of the study and ends on day 70 ±2 days. In period 2, the observation period starts on day 120 ±2 days and ends on day 140 ±2 days.
  The difference between CGM and self-monitoring of blood glucose in time below range (glucose value < 3.9 mmol/L) measured by CGM.
Time below range (glucose 3.0-3.8 mmol/L, hypoglycaemia level 1) | In period 1, the observation period begins on day 50 ±2 days of the study and ends on day 70 ±2 days. In period 2, the observation period starts on day 120 ±2 days and ends on day 140 ±2 days.
  The difference between CGM and self-monitoring of blood glucose in time below range (glucose value 3.0-3.8 mmol/L) measured by CGM.
Time above range (glucose >10.0 mmol/L) | In period 1, the observation period begins on day 50 ±2 days of the study and ends on day 70 ±2 days. In period 2, the observation period starts on day 120 ±2 days and ends on day 140 ±2 days.
  The difference between CGM and self-monitoring of blood glucose in time above range (glucose value >10.0 mmol/L) measured by CGM.
Time above range (glucose 10.1-13.9 mmol/L, hyperglycaemia level 1) | In period 1, the observation period begins on day 50 ±2 days of the study and ends on day 70 ±2 days. In period 2, the observation period starts on day 120 ±2 days and ends on day 140 ±2 days.
  The difference between CGM and self-monitoring of blood glucose in time above range (glucose value 10.1-13.9 mmol/L) measured by CGM.
Time above range (glucose >13.9 mmol/L, hyperglycaemia level 2) | In period 1, the observation period begins on day 50 ±2 days of the study and ends on day 70 ±2 days. In period 2, the observation period starts on day 120 ±2 days and ends on day 140 ±2 days.
  The difference between CGM and self-monitoring of blood glucose in time above range (glucose value >13.9 mmol/L) measured by CGM.
Mean glucose (mmol/L) | The last 20 ±2 days of each study period
  The difference between CGM and self-monitoring of blood glucose in mean glucose (mmol/L) measured by CGM.
Mean amplitude of glycemic excursions [MAGE] | In period 1, the observation period begins on day 50 ±2 days of the study and ends on day 70 ±2 days. In period 2, the observation period starts on day 120 ±2 days and ends on day 140 ±2 days.
  The difference between CGM and self-monitoring of blood glucose in mean amplitude of glycemic excursions [MAGE] measured by CGM.
Continuous overall net glycemic action [CONGA] | In period 1, the observation period begins on day 50 ±2 days of the study and ends on day 70 ±2 days. In period 2, the observation period starts on day 120 ±2 days and ends on day 140 ±2 days.
  The difference between CGM and self-monitoring of blood glucose in continuous overall net glycemic action [CONGA] measured by CGM.
Insulin dose (unit) | The last 20 ±2 days of each study period
  The difference in the mean insulin dose between CGM and self-monitoring of blood glucose.
Quality of life (EORTC QLQ-C30) | At the end of each study period (day 70 ±2 and 140 ±2).
  Difference between CGM and self-monitoring of blood glucose in quality of life assessed by EORTC QLQ-C30 questionnaire. The questionnaire has been validated for assessment of quality of life in patients with chronic pancreatitis and is composed of single-item measures and multi-item scales with scores ranging from 0 to 100 after linear transformation of the raw score. A high score for a functional scale represents a high level of functioning, as does a high score for the global health status, while a high score for the symptom items represents a high level of symptomatology.
Patient global impression of change score (PGIC) | At the end of each study period (day 70 ±2 and 140 ±2).
  Difference between CGM and self-monitoring of blood glucose in Patient global impression of change score (PGIC). The PGIC is a self-reported measure used to assess a patient's overall perception of improvement or change in their condition over time. It uses a 7-point scale, ranging from "very much improved" to "very much worse". A score ≤3 means that the condition has improved.
Hypoglycemia awareness | At the end of each study period (day 70 ±2 and 140 ±2).
  The difference between CGM and self-monitoring of blood glucose in hypoglycemia awareness assessed by the Clarke Hypoglycemia Awareness Survey. It comprises eight questions characterizing the participant's exposure to episodes of moderate and severe hypoglycemia. It also examines the glycemic threshold for, and symptomatic responses to, hypoglycemia. A score of four or more implies impaired awareness of hypoglycemia.
Standard deviation (mmol/L) | In period 1, the observation period begins on day 50 ±2 days of the study and ends on day 70 ±2 days. In period 2, the observation period starts on day 120 ±2 days and ends on day 140 ±2 days.
  The difference between CGM and self-monitoring of blood glucose in standard deviation of mean glucose (mmol/L) measured by CGM.
Coefficient of variance (%) | In period 1, the observation period begins on day 50 ±2 days of the study and ends on day 70 ±2 days. In period 2, the observation period starts on day 120 ±2 days and ends on day 140 ±2 days.
  The difference between CGM and self-monitoring of blood glucose in coefficient of variance of mean glucose (mmol/L) measured by CGM.
HbA1c (mmol/L) | At the end of each study period (day 70 ±2 and 140 ±2).
  The difference between CGM and self-monitoring of blood glucose in HbA1c mmol/L.
HbA1c (percentage) | At the end of each study period (day 70 ±2 and 140 ±2).
  The difference between CGM and self-monitoring of blood glucose in HbA1c (percentage).

CONTACTS AND LOCATIONS:
Overall Officials: Søren S Olesen, Professor, Principal Investigator — Mech-Sense, Department of Gastroenterology, Aalborg Hospital
Locations (1):
- Department of Gastroenterology, Aalborg Hospital, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2022-05-23): https://cdn.clinicaltrials.gov/large-docs/80/NCT05550480/Prot_000.pdf